CLINICAL TRIAL: NCT00429507
Title: Phase 2 Study of 153 Sm-EDTMP Followed by Autologous Peripheral Blood Stem Cell Transplantation for Breast Cancer Patients With Bone Only Metastases
Brief Title: Sm-EDTMP and Autologous Peripheral Blood Stem Cell Transplantation for Breast Cancer Patients With Bone Only Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cytogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0349; NCI-2010-00573 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Bone Metastases
Keywords: Breast Cancer; Blood Stem Cell; Bone Metastases; Radiation Therapy; Gamma Camera; Sm-EDTMP; Samarium 153-EDTMP; Stem Cell Transplant; Autologous Peripheral Blood Stem Cell Transplantation; PBSCT; Questionnaire
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Samarium 153-EDTMP + Stem Cell Transplant (Experimental): Samarium 153-EDTMP tracer dose = 30 millicurie (mCi) by vein On Day 1. If enough study drug goes to bones, will receive a higher dose of 153 Sm-EDTMP, called a therapy dose, 7-14 days after the tracer dose. Stem Cell Transplant on Day 0, about 14-21 days after Samarium 153-EDTMP. Questionnaires taking about 15 minutes to complete.
  Interventions: Drug: 153 Sm-EDTMP; Behavioral: Questionnaire; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: 153 Sm-EDTMP — Tracer dose = 30 mCi by vein On Day 1. If enough study drug goes to bones, will receive a higher dose of 153 Sm-EDTMP, called a therapy dose, 7-14 days after the tracer dose.
  Other Names: Samarium 153-EDTMP
Behavioral: Questionnaire — Questionnaires taking about 15 minutes to complete.
  Other Names: Survey
Procedure: Stem Cell Transplant — Stem Cell Transplant on Day 0, about 14-21 days after Samarium 153-EDTMP.
  Other Names: SCT; Autologous Peripheral Blood Stem Cell Transplantation; PBSCT

SUMMARY:
Primary objectives:

- To determine the time to progression in subjects with breast cancer metastatic to bone only treated with 153Sm-EDTMP and Autologous Peripheral Blood Stem Cell Transplantation (PBSCT).

Secondary objectives:

* To determine the overall survival at one year.
* To determine the efficacy of 153Sm-EDTMP at 6 months.
* To assess pain in subjects treated with 153Sm-EDTMP.
* To determine the safety of 153Sm-EDTMP.

DETAILED DESCRIPTION:
153 Sm-EDTMP is designed to provide radiation to the bone and bone marrow. The radiation may kill cancer cells.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded. You will have a physical exam. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will have a breast exam, mammogram, and computed tomography (CT) scan. You will have a bone marrow aspirate/biopsy. To collect a bone marrow aspirate/biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow/bone is withdrawn through a large needle. Blood (about 2 teaspoons) will be drawn to check the status of the disease. You will have x-rays, a bone scan, a positron emissions tomography (PET) scan, and a bone density test. Blood (about 2 teaspoons) will be drawn to check for HIV (the virus that causes AIDS), CMV (cytomegalovirus), Hepatitis B, and Hepatitis C (viruses that can infect the liver). You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will have an echocardiogram or multiple-gated acquisition scan (MUGA). An echocardiogram uses sound waves to make pictures of your heart, which helps show how well your heart pumps blood. You will be asked to lie on your left side while a technician places a probe with gel on your chest to create images of your heart to determine the function and size. You will have a lung function test to make sure your heart and lungs are healthy. You will complete a questionnaire about the pain you are experiencing. The questionnaire will take about 15 minutes to complete. Women who are able to have children must have a negative blood (about 2 teaspoons) pregnancy test.

If you are found to be eligible to take part in this study, on Day 1 you will receive a tracer dose. A tracer dose is a small amount of the study drug used to measure how the study drug is affecting the body. Your weight will be measured. Before the tracer dose is injected, you will be given fluids through a needle in your veins starting from 2 hours before the tracer dose up to 6 hours afterwards. You will receive a small amount of 153 Sm-EDTMP, called a tracer dose, through a needle in your vein.

After the tracer dose, you will have pictures taken of your body with a gamma camera 3 times that day. These photographs will be taken immediately after the dose is injected, and then 2-3 hours and 4-6 hours later. You will need to lie flat for these imaging sessions for about 10-30 minutes each time.

On Day 2, you will have 1 picture taken of your body with the gamma camera.

If, based on the photographs taken, doctors find that the drug does not go to your bones as expected, you will be removed from the study. If you leave the study at this point, you will have return to the clinic 2 times a week for the next 4 weeks. At these visits you will have a complete physical exam, and you will be asked about any side effects you may be experiencing.

If enough of the study drug does go to your bones, you will receive a higher dose of 153 Sm-EDTMP, called a therapy dose, 7-14 days after the tracer dose.

Before the therapy dose begins, you will have a physical exam, including measurement of your vital signs. Fluids will be given through a needle in your vein beginning 2 hours before the therapy dose and continuing up to 6 hours after.

You will receive the injection of 153 Sm-EDTMP through your central line. The injection will take about 15 minutes. Afterwards, your vital signs will be measured. Blood (about 2 teaspoons) will be drawn for routine tests.

The therapy dose of 153 Sm-EDTMP is expected to destroy your body's ability to make blood cells. To restore your blood-making ability, you will be given back stem cells (blood-forming cells) that will have already been taken from your body and stored for this treatment. This is called an autologous peripheral blood stem cell transplant. You will receive the stem cells given through a needle in your vein 14-21 days after the therapy dose usually as an outpatient procedure.

Family members may not be allowed with you until radiation subsides. This will reduce their exposure to radiation. You will be given instructions on how to follow radiation safety practices.

Once the radiation subsides you will be released from the hospital, at least 2 times a week you will have a complete physical exam, and you will be asked about any side effects you are experiencing. Blood (about 2 teaspoons) will be drawn up to 3 times a week until your stem cell transplant. Your vitals signs will also be checked 2 times a week.

After the transplant, at least 2 times a week for up to two (2) weeks your blood (about 2 teaspoons) will be drawn for routine tests. You will have a physical exam and your vital signs will be checked. You will receive additional care, drugs, or blood transfusions, as needed.

You will return for follow-up visits every 3 months until the end of Year 2 and then every 6 months in Years 3 and 4. Tests may occur more often if a side effect is noticed. Any side effects that you develop will be monitored until it goes away. Some of these exams and tests may take place with your home doctor, and these records will need to be sent to the study doctor so he/she can review them for careful monitoring.

In order to check the response of the cancer to the study therapy, you will have chest x-rays, CT scans, and bone scans every 3 months for the first 2 years after transplant. These will be repeated every 6 months in years 3-4 and once a year after that, as long as your cancer does not get worse. If the breast cancer has spread to your bone marrow at the time you enter this study, bone marrow biopsies will also be done at these times to see whether the cancer is responding. You will also have a PET scan at 6 months after transplant, and more often if your physician believes it will be helpful. Mammograms and bone density exams will be done once a year.

Once a year for the 10 years after you leave the study, you will have a study visit or you will be contacted by telephone. You will be asked about your general health, hospitalization, and cancer treatments.

This is an investigational study. 153 Sm-EDTMP is FDA-approved and commercially available for bone pain control. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV breast cancer metastatic to bone and/or bone marrow only.
2. Age between 18 and 65 years.
3. Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1
4. Subjects with breast tumors with hormone receptor positive disease (ER+/PR+, ER+/PR-, or ER-/PR+) must have failed at least one hormonal-based therapy for bone only disease.
5. Subjects with breast tumors with hormone receptor negative disease must have failed at least one anthracycline and/or taxane-based therapy for bone only disease.
6. White blood cell count (WBC) >/= 3.5 x10^9/L, Hb >/= 10 g/dL, platelets >/= 100 x10^9/L.
7. Adequate pulmonary function defined as forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) (corrected for hemoglobin) >/= 50% of predicted.
8. Adequate cardiac function as evidenced by left ventricular ejection fraction (LVEF) of >/= 45%.
9. Serum total bilirubin < 2x upper limit of normal (ULN), and ALT/serum glutamate pyruvate transaminase (SGPT) < 3x ULN
10. Creatinine clearance of >/= 75 mL/min for subjects up to 50 years of age, and adjusted for age by a 10% decrease per decade for subjects of more than 50 years of age.
11. Ability to understand the study and provide informed consent.

Exclusion Criteria:

1. Any metastatic disease or history of metastatic disease other than skeletal metastases
2. Impending fracture, spinal cord compression, and/or potentially unstable compression fracture of vertebral body with possibility of cord compression.
3. Previous strontium-89 or samarium-153 treatment for any skeletal involvement.
4. Cumulative external beam radiation to > 20% of marrow volume or > 40 Gy to any single region of the spinal cord.
5. Prior radiation to the bladder or kidney, defined as radiation portals that directly include any volume of either kidney and/or the bladder.
6. Life expectancy severely limited by concomitant illness (less than 6 months).
7. Prior nephrectomy.
8. History of hemorrhagic cystitis obstructive uropathy or hydronephrosis.
9. Uncontrolled arrhythmia or symptomatic cardiac disease.
10. Current gross hematuria in urinalysis (UA) in the absence of vaginal bleeding.
11. Evidence of HIV-seropositivity.
12. Inability to stop any chemotherapy treatment for breast cancer within 3 weeks preceding high dose Samarium.
13. Use of any investigational agent within 30 days preceding enrollment.
14. Pregnant or lactating women.
15. Other current or prior malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
16. Myelodysplastic syndrome.
17. Subject weight of more than 125 kg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 7, 2007 to February 4, 2010. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Samarium 153-EDTMP + Stem Cell Transplant: Samarium 153-EDTMP tracer dose = 30 millicurie (mCi) intravenous Day 1; or with study drug to bones, receive higher therapy dose of 153 Sm-EDTMP 7-14 days after tracer dose. Stem Cell Transplant Day 0, about 14-21 days after Samarium 153-EDTMP.
Period: Overall Study
Arm/Group | Samarium 153-EDTMP + Stem Cell Transplant
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Samarium 153-EDTMP + Stem Cell Transplant
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 52 [36 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression is measured as the time from study entry to the development of disease progression.
Time Frame: 7.5 Years, Study period was March 2007 to November 2014.
Measure: Median (Full Range); unit: Days
Arm/Group | Samarium 153-EDTMP + Stem Cell Transplant
Number analyzed (Participants) | 12
Days | 317 [105 to 1339]

ADVERSE EVENTS:
Time Frame: Adverse event collection from initiation of study drug administration through Day 27 post-transplant
Arm/Group | Samarium 153-EDTMP + Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Samarium 153-EDTMP + Stem Cell Transplant (N=12)
bone pain (Musculoskeletal and connective tissue disorders) | 12
nausea (Gastrointestinal disorders) | 12
stomatitis (Gastrointestinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes